CLINICAL TRIAL: NCT05202899
Title: Effect of Sugammadex for Reversal of Rocuronium-induced Neuromuscular Block on Perioperative Management of Awake Craniotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Awake Craniotomy
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Brain Tumors
Keywords: sugammadex、awake craniotomy
MeSH Terms: conditions — Brain Neoplasms | interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex Group (Experimental): rocuronium-induced general anesthesia，use of sugammadex antagonism
  Interventions: Drug: sugammadex
- Control Group (No Intervention): general anesthesia without rocuronium

INTERVENTIONS:
Drug: sugammadex — The use of sugammadex
  Other Names: Bridion; Org 25969
  Arms: Sugammadex Group

SUMMARY:
Effect of sugammadex for reversal of rocuronium-induced neuromuscular block on Perioperative Management of awake Craniotomy

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old body mass index (BMI)≥ 18.5-23.9 kg/m2, ASA grade I ~II.

Exclusion Criteria:

* Suffering from a mental illness or preoperative communication disorder, patients with claustrophobia, breathing, circulation, neuromuscular system and kidney, and other important viscera function disorder, pregnant or lactating women, a history of malignant hyperthermia, the history of drug allergy in the process of general anesthesia and recent may not used to the interaction between rocuronium, vecuronium bromide reacts drugs (such as aminoglycoside antibiotics, Anticonvulsant, magnesium).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
awake time | 10-30 minutes
  The time between asleep and awake

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China